CLINICAL TRIAL: NCT04417400
Title: Benefits of Medicines Use Review Service in Slovenia: a Randomized Controlled Trial
Brief Title: Evaluation of Medicines Use Review in Slovenia
Acronym: SLOPUZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitja Kos (Other)
Collaborators: Comunity pharmacy Celjske lekarne (Unknown); Comunity pharmacy Gorenjske lekarne (Unknown); Comunity pharmacy Goriška lekarna Nova Gorica (Unknown); Comunity pharmacy Javni zdravstveni zavod Mariborske lekarne Maribor (Unknown); Comunity pharmacy Kraške lekarne Ilirska Bistrica (Unknown); Comunity pharmacy Lekarna Brežice (Unknown); Comunity pharmacy Lekarna Kočevje (Unknown); Comunity pharmacy Lekarna Ljubljana (Unknown); Comunity pharmacy Lekarna Ormož (Unknown); Comunity pharmacy Lekarna Sevnica (Unknown); Comunity pharmacy Lekarne Ptuj (Unknown); Comunity pharmacy Obalne lekarne Koper (Unknown); Comunity pharmacy Pomurske lekarne Murska Sobota (Unknown); Comunity pharmacy Žalske lekarne Žalec (Unknown)
Responsible Party: Sponsor-Investigator, Mitja Kos, prof. dr. Mitja Kos, Head of the Department of Social Pharmacy, University of Ljubljana
Organization: University of Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MZ 0120-321/2016-2; P1-0189 (Other Grant/Funding Number: A PhD under research group funded by Slovene Research Agency.)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Medicines Use Review Service; Multiple Medication; Adherence, Medication
Keywords: adherence; medicines use review; drug related problems; cognitive pharmaceutical service; community pharmacy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Upon enrollment patients were centrally randomized into two groups -test and control. Patients from the test group received MUR at visit 1. After 12 weeks both groups were reinterviewed. Upon study completion, patients from the control group received MUR due to ethical reasons, however the documentation was not part of the study anymore.
Masking Description: Patients and pharmacist were blind to the intervention at the time of enrollment.
  Afterwards, pharmacist were notified about the randomization to be able to prepare for the patients that will receive MUR at the visit 1. Patients were blinded until the visit 1 - until after the baseline data collection"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients who received MUR at visit 1
  Interventions: Behavioral: medicines use review
- Control (No Intervention): Patients received standard care and MUR after visit 2 (upon completion of the study)

INTERVENTIONS:
Behavioral: medicines use review — The provision of MUR service as defined in the SOP MUR (Slovene Chamber of Pharmacies). It is classified as a type 2a review (PCNE typology) and it is intended for the patients to support them in regular and proper medicines use. MUR is performed based on medication history and information provided by the patient in a purposely scheduled conversation with the pharmacist. Pharmacists must be certified to provide MUR. MUR goal is to identify DRPs and recommend interventions to resolve them. During the MUR interview, the pharmacist completes a working sheet that records information regarding medicines, identified DRPs and recommended interventions. After the MUR interview, patients are provided with a personal medicines card that contains all the information that is needed to support effective and safe medicines use (dosing regimen, taking with/without food, special warnings, recommendations, etc.).
  Arms: Intervention

SUMMARY:
Medicines Use Review service (PUZ) has been officially introduced in Slovenian pharmacy practice in 2015 and has been offered to pharmacy customers by pharmacist, certified to provide the service. Patients can to talk to a pharmacist and discuss their medicines, how they use it and any issues or question they might have. We designed a study to evaluate how Medicines Use Review (PUZ) work and how it is reaching the set objectives. The objectives of the PUZ service are to address actual patient medicines use and consequently improve medication adherence, identify and solve drug related problems and enhance medication knowledge. Pharmacists, who are certified to provide the service, recognized the patients, who might need the service and invited them to participate in the study. The study consisted of two visits in 12 weeks' time period. Patients, who decided to participate, were randomly allocated in two groups - intervention and control. Both groups were interviewed and fulfilled questionnaires at visit 1 (V1). Afterwards the test group patients received PUZ. After 12 weeks both groups attended the visit 2 (V2), where they were re-interviewed and fulfilled questionnaires again. After the study completion also the patients from control group received PUZ due to ethical reasons.

ELIGIBILITY:
Inclusion Criteria:

* at least one prescription medicine for a chronic condition for at least six months
* deemed to be suitable for MUR by a pharmacist, certified to provide the MUR service;
* ability to communicate in Slovenian; The inclusion of patients was performed in accordance with the SOP MUR, to reflect how patients are generally offered MUR service in Slovenia.

Exclusion Criteria:

* urgent need of MUR (the service delay due to randomization would risk their health);
* referred for MUR by a healthcare professional (general practitioner, nurse, etc.);
* the patient's carer, rather than the patient themselves, was able to attend the interviews and receive MUR;
* previously received MUR or an advanced medication review;
* difficulties understanding, communicating or other issues (vision, hearing) that might affect study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
medication adherence | 12 weeks (V2-V1)
  Self-reported medication adherence to multiple medications, evaluated by an 8-item Morisky Medication Adherence Scale (©MMAS-8) and scored with ©Morisky Widget MMAS-8 Software. MUR impact was defined as the relative difference in in MMAS-8 score after 12 weeks (V2-V1) between test and control group.

SECONDARY OUTCOMES:
drug-related problems | 12 weeks (V2-V1)
  The changes in the proportion of manifested DRPs, the proportion of patients with at least one mDRPs, and the risk of the mDRPs between visits. This outcome only considered for the intervention group (test group), therefore the before-after analysis was applied.
Medicine-associated burden | 12 weeks (V1-V2)
  MUR impact on medicine-associated burden was defined as the mean relative difference in the score of Living with Medicines Questionnaire (©LMQ), visual analog scale (VAS) and each domain score between test and control group after 12 weeks (V1-V2).
Patient information ('knowledge') regarding medicines | 12 weeks
  Interview with the patients. Patients answered three questions regarding each of their regularly used prescription medicines: (i) "What are you taking the medicine for?", to state the purpose of medicine use; (ii) "How are you supposed to take the medicine?", to state the daily dose; and (iii) "Do you know of any special warnings regarding the medicine? If yes, which ones?". Accuracy of answers regarding the purpose of medicine and its daily dose were checked by comparing them with either physician instructions or, when physician instructions were unavailable, Summary of Product Characteristics (SmPC). Answers were deemed to be 'correct' if they matched the information in these sources, 'incorrect' if they did not match or 'not known' if patients responded with "I don't know" or 'no'. Proportions of correct and incorrect answers per patient-medicine, and proportions of improvement or deterioration in given information between visits for the test and control group, were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Locatelli, M.Pharm, PhD, Study Director — University of Ljubljana; Mitja Kos, MPharm, PhD, Principal Investigator — University of Ljubljana; Urska Nabergoj Makovec, MPharm, Study Chair — University of Ljubljana
Locations (14):
- Slovenia (14):
  - Community pharmacy "Lekarna Brežice", Brežice
  - Community pharmacy "Celjske lekarne javni zavod", Celje
  - Community pharmacy "Kraške lekarne Ilirska Bistrica", Ilirska Bistrica
  - Community pharmacy "Lekarna Kočevje", Kočevje
  - Community pharmacy "Obalne lekarne Koper", Koper
  - Community pharmacy " Gorenjske lekarne", Kranj
  - Community pharmacy "Lekarna Ljubljana", Ljubljana
  - Community pharmacy "Javni zdravstveni zavod Mariborske lekarne Maribor", Maribor
  - Community pharmacy "Pomurske lekarne Murska Sobota", Murska Sobota
  - Community pharmacy "Goriška lekarna Nova Gorica", Nova Gorica
  - Community pharmacy "Lekarna Ormož", Ormož
  - Community pharmacy "Lekarne Ptuj", Ptuj
  - Community pharmacy "Lekarna Sevnica", Sevnica
  - Community pharmacy "Žalske lekarne Žalec", Žalec

IPD SHARING:
Plan to Share IPD: No
We plan to publish the results of the study in a form of original research manuscript in an international journal with the impact factor. Any questions regarding the study protocol, process and analysis can be address to the principal investigator.

REFERENCES:
- [Background] Nabergoj Makovec U, Kos M, Pisk N. Community pharmacists' perspectives on implementation of Medicines Use Review in Slovenia. Int J Clin Pharm. 2018 Oct;40(5):1180-1188. doi: 10.1007/s11096-018-0644-6. Epub 2018 Jun 16. PMID 29909563
- [Background] Griese-Mammen N, Hersberger KE, Messerli M, Leikola S, Horvat N, van Mil JWF, Kos M. PCNE definition of medication review: reaching agreement. Int J Clin Pharm. 2018 Oct;40(5):1199-1208. doi: 10.1007/s11096-018-0696-7. Epub 2018 Aug 2. PMID 30073611
- [Derived] Nabergoj Makovec U, Locatelli I, Kos M. Improved adherence with Medicines Use Review service in Slovenia: a randomized controlled trial. BMC Health Serv Res. 2021 Mar 22;21(1):266. doi: 10.1186/s12913-021-06223-8. PMID 33752647